CLINICAL TRIAL: NCT07230704
Title: Effects of Low-Flow and Standard-Flow Sevoflurane Anesthesia on Perioperative Inflammation in Bariatric Surgery
Brief Title: Effects of Low-Flow and Standard-Flow Sevoflurane Anesthesia on Inflammatory Markers in Bariatric Surgery
Acronym: LOWBAR
Status: Completed | Type: Observational
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Uğur serkan Çitilcioğlu, Principal Investigator, Department of Anesthesiology, Adana City Training and Research Hospital
Other Study IDs: ADN-LOWFLOW-2025; 10-354 (Other: Adana City Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Inflammation; Bariatric Surgery Candidate
Keywords: Sevoflurane; Low-Flow Anesthesia; Inflammatory Markers; Hemodynamics
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-flow Sevoflurane: Patients who underwent laparoscopic sleeve gastrectomy under general anesthesia with low-flow sevoflurane (fresh gas flow = 1 L/min). Data were obtained retrospectively from hospital records.
- Standard-flow Sevoflurane: Patients who underwent laparoscopic sleeve gastrectomy under general anesthesia with standard-flow sevoflurane (fresh gas flow = 4 L/min). Data were obtained retrospectively from hospital records.

SUMMARY:
This retrospective observational study aimed to compare the effects of low-flow and standard-flow sevoflurane anesthesia on perioperative inflammatory responses in patients undergoing laparoscopic sleeve gastrectomy for obesity. Data were obtained from the anesthesia and laboratory records of 155 adult patients who received either low-flow (1 L/min) or standard-flow (4 L/min) sevoflurane anesthesia between January 2022 and January 2025 at Adana City Training and Research Hospital. Preoperative and postoperative inflammatory markers, including C-reactive protein (CRP), neutrophil-to-lymphocyte ratio (NLR), and red cell distribution width (RDW), were recorded and compared between the two groups. Hemodynamic parameters such as mean arterial pressure and heart rate were also analyzed to assess intraoperative stability. The primary objective of the study was to evaluate the impact of anesthetic flow rate on perioperative inflammation, while the secondary objective was to assess hemodynamic stability during anesthesia. This study may contribute to a better understanding of how low-flow anesthesia influences systemic inflammatory responses and perioperative hemodynamics in morbidly obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
This retrospective observational cohort study investigated the effects of low-flow and standard-flow sevoflurane anesthesia on perioperative inflammatory markers and hemodynamic stability in patients with obesity undergoing laparoscopic sleeve gastrectomy. The study included 155 adult patients operated between January 2022 and January 2025 at Adana City Training and Research Hospital, Adana, Turkey.

Patients were divided into two groups according to the fresh-gas flow rate used during anesthesia:

Low-flow group: sevoflurane with a total fresh-gas flow rate of 1 L/min,

Standard-flow group: sevoflurane with a total fresh-gas flow rate of 4 L/min.

All patients received general anesthesia as part of routine clinical care. No randomization or intervention was performed by the investigators. Demographic characteristics, anesthesia records, intraoperative hemodynamic parameters (mean arterial pressure, heart rate), and perioperative laboratory results were obtained retrospectively from hospital electronic records.

Preoperative and postoperative (24-hour) values of inflammatory markers-including C-reactive protein (CRP), neutrophil-to-lymphocyte ratio (NLR), and red cell distribution width (RDW)-were compared within and between groups. The primary endpoint was the change in these inflammatory biomarkers between pre- and postoperative measurements. The secondary endpoint was the comparison of intraoperative hemodynamic stability (MAP and HR variability, incidence of hypotension or bradycardia) between the two groups.

This study aims to provide evidence regarding whether low-flow sevoflurane anesthesia (1 L/min) offers comparable or superior inflammatory and hemodynamic profiles compared with standard-flow anesthesia (4 L/min) in morbidly obese patients. The findings may help optimize anesthetic techniques for bariatric surgery by balancing patient safety, hemodynamic stability, and environmental considerations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years
* Underwent laparoscopic sleeve gastrectomy under general anesthesia
* Received low-flow or standard-flow sevoflurane anesthesia
* ASA physical status I-III
* Complete perioperative records available

Exclusion Criteria:

* Conversion to open surgery
* Incomplete or missing data
* Significant comorbidities (e.g., severe cardiac, hepatic, or renal dysfunction)
* Perioperative complications unrelated to anesthesia
* Age <18 or >60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Retrospective analysis of 155 adult patients who underwent laparoscopic sleeve gastrectomy under general anesthesia between January 2022 and January 2025 at Adana City Training and Research Hospital. Patients were grouped according to the fresh gas flow rate used during anesthesia (low-flow vs. standard-flow sevoflurane).
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in C-reactive protein (CRP) concentration | From preoperative baseline to postoperative 24 hours
  Change in serum C-reactive protein (CRP) levels from preoperative baseline to postoperative 24 hours will be compared between low-flow and standard-flow sevoflurane groups.
Change in neutrophil-to-lymphocyte ratio (NLR) | From preoperative baseline to postoperative 24 hours
  Change in neutrophil-to-lymphocyte ratio (NLR) from preoperative baseline to postoperative 24 hours will be compared between low-flow and standard-flow sevoflurane groups.
Change in red cell distribution width (RDW) | From preoperative baseline to postoperative 24 hours
  Change in red cell distribution width (RDW) from preoperative baseline to postoperative 24 hours will be compared between low-flow and standard-flow sevoflurane groups.

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) variability | From induction of anesthesia to end of anesthesia
  Change and variability in intraoperative mean arterial pressure (MAP) recorded throughout anesthesia will be compared between low-flow and standard-flow sevoflurane groups.
Heart rate (HR) variability | From induction of anesthesia to end of anesthesia
  Change and variability in intraoperative heart rate (HR) recorded throughout anesthesia will be compared between low-flow and standard-flow sevoflurane groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur serkan Citilcioglu, MD, Principal Investigator — Adana City Training and Research Hospital
Locations (1):
- Adana City Training and Research Hospital, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to institutional data protection policies.